CLINICAL TRIAL: NCT05954923
Title: The Glucagonotropic Effect of Amino Acids in Humans
Acronym: STAMINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Malte Palm Suppli, MD, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STAMINA
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, single-arm study. Participants act as their own controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary arm (Experimental): This is a single-arm study. Each subject will participate in 6 experimental days in a randomized order. The interventions are equimolar bolus infusions of A) glutamine, B) arginine, C) alanine, D) leucine, E) proline and F) saline (placebo)
  Interventions: Other: Amino acid bolus infusion

INTERVENTIONS:
Other: Amino acid bolus infusion — Equimolar bolus infusions of amino acids or saline (placebo)

SUMMARY:
The objective of the study is to delineate the glucagonotropic signal exerted by selected amino acids in human subjects as well as the metabolic clearance rate of these amino acids after intravenous infusion

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, each participant giving written informed consent will participate in six experimental days. The glucagonotropic effect and metabolic clearance of selected amino acids and saline (placebo), respectively, will be evaluated in 12 healthy individuals. After screening, each participant will undergo 6 double-blinded experimental days performed in randomized order. The experimental days will each last 75 minutes. The amino acids selected for the experiment are glutamine, arginine, alanine, leucine and proline.

ELIGIBILITY:
Inclusion Criteria:

* normal fasting plasma glucose and glycated hemoglobin (HbA1c) < 42 mmol/mol
* body mass index (BMI) between 18.5 and 25 kg/m2
* Hemoglobin > 8.3 mmol/L
* Age between 20 and 65 years
* oral and written informed consent

Exclusion Criteria:

* Diabetes
* first-degree relatives with diabetes
* fasting plasma triglycerides indicating dyslipidemia (> 2 mmol/L)
* nephropathy (eGFR < 60 ml/min) and/or microalbuminuria (albumine/creatinine ratio > 30 microgram/mg)
* liver disease and/or ALT and/or AST levels > 2 x upper normal reference limits.
* signs of liver fibrosis and/or steatosis evaluated by transient elastography (CAP > 238 dB/min) and/or kPa > 6.0) and/or FIB-4 index > 1.45
* regular use of prescription medication
* use of dietary protein supplementation
* any condition the investigator feels would interfere with trial completion

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
bsAUC30 | bsAUC is calculated from blood samples drawn at times 0 min, 1 min, 2 min, 4 min, 6 min, 10 min, 15 min and 30 min
  Baseline subtracted area under the curve for glucagon concentration during the first 30 minutes of the experiment

SECONDARY OUTCOMES:
AUC30 | AUC30 is calculated from blood samples drawn at times 0 min, 1 min, 2 min, 4 min, 6 min, 10 min, 15 min and 30 min
  total area under the curve for glucagon concentration during the first 30 minutes of the experiment
AUC60 | AUC60 is calculated from blood samples drawn at times 0 min, 1 min, 2 min, 4 min, 6 min, 10 min, 15 min, 30 min and 60 min
  total area under the curve for glucagon concentration the first 60 minutes of the experiment
bsAUC60 | bsAUC60 is calculated from blood samples drawn at times 0 min, 1 min, 2 min, 4 min, 6 min, 10 min, 15 min, 30 min and 60 min
  Baseline subtracted area under the curve for glucagon concentration during the first 60 minutes of the experiment
peak glucagon concentration | measured between time 0 min and time 60 min
  the highest concentration of glucagon after infusion of amino acids/placebo

OTHER OUTCOMES:
Metabolic clearance of amino acids | Time 0 min to time 60 min
  The metabolic clearance of each infused amino acid calculated from amino acid concentrations
Insulin | Time -15 min to time 60 min
  plasma concentration of insulin during the experiment
C-peptide | Time -15 min to time 60 min
  plasma concentration of C-peptide during the experiment
Total and individual amino acids | Time -15 min to time 60 min
  plasma concentration of total and individual amino acids during the experiment
GLP-1 | Time -15 min to time 60 min
  plasma concentration of glucagon-like peptide 1 (GLP-1) during the experiment
GIP | Time -15 min to time 60 min
  plasma concentration of glucose-dependent insulinotropic polypeptide (GIP) during the experiment

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All published data will be made available to other researchers upon reasonable request